CLINICAL TRIAL: NCT01910428
Title: A Phase I Study of L-asparaginase Encapsulated in Red Blood Cells (Eryaspase) in Combination With the CALGB Regimen During Induction and Consolidation Phases in the Treatment of Adult Patients With Acute Lymphoblastic Leukemia and Lymphoma
Brief Title: L-asparaginase Encapsulated in Red Blood Cells (Eryaspase) for Treatment of Adult Patients With ALL or LBL
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor decision based off site/PI feedback about
Sponsor: ERYtech Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GRASPALL 2012-09
Record Dates: First submitted 2013-07-24; First posted 2013-07-29 (Estimated); Last update posted 2018-07-05 (Actual); Status verified 2018-07

CONDITIONS: Acute Lymphoblastic Leukemia; Lymphoblastic Lymphoma
Keywords: L-asparaginase encapsulated in RBCs, leukemia, lymphoma
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia; Lymphoma | interventions — Erythrocyte Count; eryaspase

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- L-asparaginase encapsulated in RBC (Experimental): L-asparaginase encapsulated in RBC dose titration: 50, 100, 150 or 200 IU/kg
  Interventions: Drug: L-asparaginase encapsulated in RBC

INTERVENTIONS:
Drug: L-asparaginase encapsulated in RBC — * 50 IU/kg IV
  * 100 IU/kg IV
  * 150 IU/kg IV
  * 200 IU/kg IV
  Other Names: ERYASPASE

SUMMARY:
Asparaginase (Asp) is used during the induction phase of ALL treatment for children and young adults. Its efficacy is counterbalanced by its toxicity, mainly in patients 40 years or older. The efficacy rate in older adult population is lower than for children or young adults. A recent review on outcomes in older adults with ALL pointed out that there were significantly more drug reductions, omissions or delays in the older group as compared to younger adults and that asparaginase was the drug most commonly omitted.

The investigational product ERYASPASE is a dispersion for infusion of homologous red blood cells (RBC) encapsulating E. coli L-asparaginase.

A previous European phase I/II clinical study in children and adults (<55 yo) at first relapse of ALL was conducted to determine the optimal dose of homologous RBC encapsulating native E. coli Asp (GRASPA®) in 24 patients with relapsed ALL. The activity and safety profiles of 3 doses of GRASPA® (50, 100 and 150 IU/kg) in combination with standard chemotherapy were compared to free native Asp. The global safety profile is also improved, reducing hypersensitivity, liver toxicity and coagulation disorders. Study showed that a single dose of GRASPA® 150 IU/kg induced a depletion in plasmatic asparagine for 18.6 days, i.e. similar to that obtained with 8 injections of 10,000 IU/m² of free native Asp. A reduction in the incidence and severity of the allergic reactions and coagulation disorders were observed with GRASPA® (Domenech 2011).

A French phase II study designed to determine the maximum tolerated dose of GRASPA® in combination with a polychemotherapy regimen in ALL patients older than 55 yo at first diagnosis has been performed, and showed that both 100 and 150 IU/kg doses fulfilled the predefined criteria for efficacy and tolerability but the better profile of 100 IU/kg dose was considered the optimal dose in this setting. A phase II/III trial in adult and children patients with relapsed ALL is currently ongoing.

Based on these results, the combination of ERYASPASE with the CALGB chemotherapy regimen appears to be an attractive combination for the treatment of adults patients with ALL/LBL.

DETAILED DESCRIPTION:
A phase I study to assess the limiting toxicities, global safety and clinical activity of ERYASPASE, using a dose titration design to confirm that the safety profile of ERYASPASE in combination with the CALGB chemotherapy regimen is similar to that observed in the European chemotherapy regimen. PK/PD and immunogenicity parameters will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 18 years and over
* Diagnosis of acute lymphoblastic leukemia or lymphoblastic lymphoma
* Received no more than 1 prior treatment for ALL/LBL
* Note: Patients who have received transplant during 1st remission are excluded since this would be considered a 2nd treatment
* ECOG performance status 0-2
* Signed Informed Consent Form

Exclusion Criteria:

* Other serious medical illness other than that treated by this study which would limit survival to <2 years or psychiatric conditions which would prevent informed consent or compliance with treatment.
* Presenting with a general or visceral contraindication to intensive treatment including:

  * uncontrolled or severe cardiovascular disease, including recent (<6 months) myocardial infarction or congestive heart failure,
  * Current Grade 3 or higher coagulopathy, thrombosis and/or hemostasis disorders,
  * Serum creatinine concentration, 1.5 times greater than the upper limit of laboratory normal ranges (ULN), except if related to ALL/LBL,
  * total bilirubin 1.5 times greater than the ULN, except if related to ALL/LBL,
  * transaminases (AST or ALT) levels, 5 times greater than the ULN, except if related to ALL/LBL,
  * An uncontrolled bacterial, viral, or fungal infection or an active duodenal ulcer, until these conditions are corrected or controlled.
* History of Grade 3 or higher allergic reaction with prior asparaginase treatment,
* History of allergy to penicillin or related antibiotic
* History of Grade 3 or higher blood transfusion incident according to US Biovigilance Network which refers to any transfusion followed by a major intervention (vasopressors, intubation, transfer to intensive care) to prevent death.
* Presenting with anti-erythrocyte antibodies leading to the unavailability of phenotype compatible red blood cells.
* Participation in a clinical study involving receipt of an investigational drug during the last 30 days.
* Women of childbearing potential without effective contraception as well as pregnant or breast feeding women.
* Patient receiving treatment likely to cause hemolysis or under phenytoin treatment.
* Patient undergoing yellow fever vaccination.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2013-10 (Actual); Primary Completion 2018-01-25 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Determination of the Maximal Total Dosage (MTD) based on number of patients presenting with related DLT | Duration of study
  ERYASPASE administered during the induction and consolidation phases of the standard multi-agent CALBG chemotherapy

SECONDARY OUTCOMES:
Overall safety and tolerability | Duration of study
  Number, incidence, type, severity, outcome and causality of AE and SAE
Plasma concentrations of asparagine,aspartate,glutamine and glutamate. | Induction and consolidation phases
  Pharmacodynamic parameters (PD)
Optional samples for CSF levels of amino acids | Induction and consolidation phases
  PD parameters
Red blood cell 24-hour recovery analysis , total, free and encapsulated L-asparaginase | Day of administration and 24h post administration
  Pharmacokinetic parameter
Immunogenicity | Duration of study
  Evaluation of the titer of the anti-asparaginase antibody

OTHER OUTCOMES:
Response to treatment | Induction and consolidation phases
  Hematological Complete Response rate

CONTACTS AND LOCATIONS:
Overall Officials: Richard A LARSON, MD, Principal Investigator — University of Chicago
Locations (5):
- United States (5):
  - University of Chicago, Chicago, Illinois
  - University of Maryland, Greenebaum Comprehensive Cancer Center, Baltimore, Maryland
  - Monter Cancer Center, Lake Success, New York
  - Duke University, Durham, North Carolina
  - Ohio State University, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: Undecided